CLINICAL TRIAL: NCT03952741
Title: Cognitive Functional Therapy (CFT) Compared to Cognitive Patient Education and Physiotherapy (COPE-PT) for Patients With Non-specific Chronic Low Back Pain (NSCLBP)
Brief Title: Cognitive Functional Therapy Compared to Cognitive Patient Education and Physiotherapy for Patients With Low Back Pain
Acronym: FAktA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Kjartan Vibe Fersum, Associate Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 250.05
Record Dates: First submitted 2017-11-13; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Functional Therapy (Experimental): The intervention is a targeted cognitive functional therapy and will be based on examination findings. It is behaviorally directed with a focus on normalizing mal-adaptive pain, cognitive and movement behaviors in a graduated manner. In the evaluation process it is considered whether the patient has adjusted to the back complaints in a positive way (confrontation, active coping, minimal avoidance behavior) or in a negative way (passive coping, fear and avoidance behavior). Work related issues will be a particular focus, with the aim of achieving close co-operation between the worker, the workplace and the worker's responsible health care provider.
  Interventions: Behavioral: Physical Therapy
- Cognitive Patient Education and PT (Active Comparator): The intervention in the second group will receive much training in cognitive coping techniques after the COPE LBP trial principles (Werner et al. 2010). The educational part of the COPE for new instructors with a PT background takes 2 days supervised by Werner and his group, with regular follow-up meeting with the project leaders, together with a psychologist trained in cognitive therapy
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Physical Therapy
  Other Names: Cognitive functional therapy and Cognitive patient education

SUMMARY:
Background: There is a need for projects that link work closer to the rehabilitation chain to further understand risk factors for sick-leave. The new aspect of this project is that it combines work place intervention with individualized physiotherapy, based on validated standardized tests and a classification based treatment system.

Aim: The aim is to expand the knowledge and understanding of complex causes of musculoskeletal pain, particularly low back pain (LBP). The main aim is to examine if cognitive functional therapy (CFT) can further reduce sick-leave and pain, and increase function and well-being.

Material and methods: To ensure good recruitment we have collaboration with the Department for Health and social services in the county of Bergen, which has a sickness absence above average among their health workers.

We will invite those with LBP problems to be included in an RCT and receive CFT in a physiotherapy clinic (usually offered 5 to 12 visits). The comparison group will receive a series with cognitive patient education and physiotherapy (COPE-PT) given by a physiotherapist. All participants will be followed by their workplace leaders. All patients who enter the RCT will be re-examined at 3 and 12 months and the predictors for sick-leave, function and coping in different sub-groups of patients with NSLBP will be studied.

DETAILED DESCRIPTION:
Musculoskeletal complaints: Function, activity and work

1. Introduction and relevance

Causes of sick-leave are multidimensional, and even if a sick-listed person has physical pain and/or functional problems, treatment models that focus only on these aspects are often not successful. In fact a sole focus on physical impairment may even medicalize the problem and increase a person's dependency on care professionals. Current knowledge suggests it is necessary to combine cognitive, functional and organizational strategies which include the workplace leader in order to reduce sick-leave absence. High quality clinical studies set in a Norwegian workplace that take all these aspects into consideration are scarce, and there is a need for research in which multiple dimensions are integrated in the management of persons who are, or are about to become sick-listed.

Musculoskeletal complaints and particularly non-specific low back pain (NSLBP) is a common reason for sick-leave in Norway. Risk profiling and stratification of workers with NSLBP is central in this project. Differences in functional capacity and requirements, particularly at work and in activities of daily living, means that workers with similar medical diagnoses may need different treatments. This research project proposes a several stages process. In the first stage, those workers who become sick-listed, or who are on the brink of becoming so, due to musculoskeletal complaints, including NSLBP, will be closely supported by specially trained workplace leaders with a focus on preventing medicalization of the problem and promoting activity. It is a legal responsibility for every workplace in Norway to take care of workers with health problems, but this has in many work-places not been optimized. In the next stage those who have musculoskeletal complaints will be invited to undergo a functional evaluation 4 weeks after their first day of sick-leave or start of their complaint. This functional evaluation can be used in the communication between the patient, their work leader and/or their primary health caretaker. Those with LBP will be invited to test an intervention model that builds on recent knowledge about sub-classification of NSLBP to reduce sick-leave, improve function and coping. This treatment is called cognitive functional therapy (CFT), will be tested in a randomized, controlled trial (RCT). There will be a comparison group in the RCT who will get a series with cognitive patient education and physiotherapy (COPE-PT) by specially trained physiotherapists. All participants will be followed by their work leaders. To enhance understanding about the causes and mechanisms of sick-leave, and to understand workers experience of treatments as well as the work leaders experience of the educational courses and their use of the functional evaluation, a parallel qualitative process evaluation will take place. The project intends to increase our knowledge of risk factors for sickness absence and how to improve the communication between the patient, their workplace and caretakers.

2 Stratification of back pain has received increased attention the last few years. There is increasing evidence that interventions based on a multidimensional understanding of patients with back- and pelvic related problems allowing more targeted intervention and can have implications for the treatment effect (Main & Watson 1996; O'Sullivan 1997; Linton 2000; Skouen et al. 2002; Fritz et al. 2003; Fersum et al. 2009). It is important that the multidimensional intervention takes place within a bio-psycho-social perspective, enabling targeted intervention towards the underlying mechanisms of pain and disability.

Cognitive patient education (COPE) for patients with musculoskeletal pain problems, including LBP, has for the last few years become an element, either alone or as part of multidisciplinary pain programs (Moseley et al. 2004; Werner et al 2010).

3. Methods and material

This study is a RCT for patients with NSLBP. Those with remaining LBP complaints at this stage will be randomized to either targeted cognitive functional therapy (CFT) intervention taking place in a physiotherapy clinic or to a comparison group with cognitive patient education and physiotherapy (COPE-PT). All will be followed by their workplace leader at their individual workplace.

Research questions:

RCT study: Persons with 4-8 weeks of sick-leave and/or who has remaining NSLBP at this stage: Do workers receiving cognitive functional therapy (CFT) combined with workplace intervention, have reduced sick-leave, improved function and coping, compared to those receiving cognitive patient education and physiotherapy (COPE-PT), in combination with workplace intervention, at 3 and 12 months after the intervention?

Material, design and outcome measures

Study

Cognitive functional therapy (CFT) compared to cognitive patient education and physiotherapy (COPE-PT) for patients with non-specific chronic low back pain (NSCLBP):

Participants with NSCLBP will be recruited as part of another study related to the FAkta project. Before randomization all patients will be examined with standardized tests as well as with a short walking test with the use of an accelerometer.

Workers with NSLBP will be randomized to either CFT (O'Sullivan, 2000, 2005) or to a comparison group with COPE-PT. All participants will be followed by their workplace leaders. Persons who randomly are allocated to either the CFT intervention group or comparison group COPE-PT will be offered treatment by specially trained physiotherapists at a physiotherapy clinic, based on the multidimensional understanding of their complaints.

Outcome measures: The primary outcome measure in the RCT is sick-leave, measured by number of days absence from work. The participants in this study will, in addition to the questionnaires mentioned above, have the the Roland Morris questionnaire as secondary outcome measure. The project will start at the beginning of 2012, and persons will be included until the end of 2013, with the last follow-up at the end of 2014.

Power calculation: In a former study (Steenstra et al. 2006) where a similar model for workplace intervention was evaluated, an average of 100 days (SD=96.0) of sick-leave was found for back patients who received intervention, compared to 130 days (SD=70.0) in those who received treatment-as-usual. A sample size of 123 participants in each group gives a power of 80 % to detect an effect of this magnitude with significance level at 0.05.

However, a recent power calculation based on the recent results from Fersum et al. (2013) where CFT was compared to manual therapy indicate that it should be sufficient with 30 participants in each group. The results have still not been published internationally, but measured in effect size (ES), the difference between the new CFT compared to today's usual practice with manual therapy and exercise was around 1 ES on most measures, in favor of the CB-CFT, reflecting both a statistical and clinical significant difference. The participant in this new study will, however, probably have more problems compared to the previous RCT. This has enabled us to aim for intervention group and one comparison group with at least 50, but hopefully close to 70 in each group. This sample size will give adequate power to detect sick-leave differences of this magnitude, even allowing for a substantial attrition rate.

Personal resources in the study : All PTs that will take part in study will receive an instructional course covering subjects like work life, optimal cognitive approach for the patients, and strategies to ensure optimal co-operation between the workplace and the worker. Three of these experienced therapists will have specialized training in the CFT intervention, which they have already utilized in participation in a similar, recent RCT. The 4-5 PTs in the second intervention group will not be familiar with CFT, but they will receive much training in cognitive coping techniques after the COPE-PT LBP trial principles (Werner et al. 2010). The educational part of the COPE-PT for new instructors with a PT background takes 2 days supervised by Werner and his group, with regular follow-up meeting with the project leaders, together with a psychologist trained in cognitive therapy (Minna Hynninen).

The CFT is adjusted to the individual, with minimum duration of 45 minutes each session, and 4 - 8 treatments during a period of 8 - 12 weeks (average 7-8 treatments). Follow-up will take place after the intervention period (at 3 months) and will include a physical examination and questionnaires. The next follow-up will be at 12 months and by questionnaires only. The participants in COPE-PT will receive one weekly session 4 times, and the follow-up examination will also be at 3 and 12 months, similar to the CFT group.

The person in charge of the RCT is researcher Kjartan Vibe Fersum, who will assist in the project co-ordination and CFT treatment. Alice Kvåle will together with the research fellow Tove Ask be an assessor of all patients who enter the project at 4-6 weeks. Only Kvåle will do the re-examination at 3 months of patients who have entered the RCT and she will be blinded for group belonging.

4. Organization, budget and relevance

Project management, organisation and cooperation The Physiotherapy research group, unit for Musculoskeletal complaints, at the Department of Public Health and Primary Health Care, University of Bergen (UiB) is responsible for managing and organizing the project, in cooperation with the Department of Health- and Social Services at Bergen County. This department has documented above average sick-leave among their health service employees, and both the management and the political leaders of the department aim to reduce this.

Budget This project has got Nkr. 4.700.000,- from the Norwegian Fund for Postgraduate Training in Physiotherapy to cover expenses for Kjartan Vibe Fersum and Tove Ask in the time period 2011 to 2015. Other resources are either part of our research positions at UiB or have been/will be applied for. Details are found in Appendix IV. The Department of Health and Social Services at Bergen County has agreed to let the workplace leaders and union leaders have paid leave when participating in the education courses and/or in the focus group interviews.

Compliance with strategic documents At the Department of Public Health and Primary Health Care, UiB, we have many resource persons who have musculoskeletal pain as their major area of interest, which is reflected both in the departments' research and teaching. One major goal is to further enhance knowledge and understanding regarding the complex causes and mechanisms of musculoskeletal pain and disability, as well as to examine the effect of a targeted functional approach in combination with focus on the workplace, evaluated both on the individual and the societal level. Part of this project aims to identify subgroups of workers with non-specific low back pain who just have been sick-listed or who are about to be so. This allows workers to be classified in such a way that they will respond to targeted treatment and get substantial improved effect of the intervention in comparison to what is usual today. The project will be performed in close co-operation with the Department of Health and Social Services, Bergen County.

Relevance to society In a recent reform for interaction between the municipalities and secondary health services in Norway ("Samhandlingsreformen" 2010), the importance of increased focus on health promotion and rehabilitation within the local councils has been underlined. A more efficient system of management and treatment within the primary health care system should prevent more extensive and chronic complaints. Recognition of the early signs and risk factors of musculoskeletal complaints in a bio-psycho-social perspective in different subgroups of workers is of great importance. Health promotion and rehabilitative measures must recognize the different needs of different groups ("Rett behandling, på rett sted, til rett tid" - Jfr. St.m.47). Effective communication between the worker, the workplace and the treating PTs/MTs in the municipality are central. The workers who are recruited to the project are themselves all workers within the Department of Health and Social Services. Their work is often quite physically demanding, and they have an above average percentage of sick-leave. It is challenging to try to improve function in workers with heavy workloads in order to reduce sick-leave, for the benefit of the individual and for society.

The project is likely to have important consequences regarding how workers at risk are cared for in the workplace, potentially highlighting the need for the right actions to the right time. The results of this study may lead to better interaction between health personnel (here mainly PTs/MTs), the work place and the occupational health services. The RCT will clarify whether classification based CFT results in greater improvements in function and working ability, than treatment-as-usual. The qualitative part of the project will give insight into the mechanisms for sick-leave, and give additional information as far as aspects that can be improved in to enhance workplaces effectiveness in dealing with musculoskeletal complaints, especially with reference to workers with back problems.

Environmental perspectives By means of the RCT the aim is to test if the new treatment model of CFT combined with focus on the workplace, will lead to improved function and less sickness absence, in comparison to a cognitive treatment strategy without hands-on.

5. Ethics

Ethical aspects There is no harm related to participation in the project. The participants will get written and verbal information about the project via their workplace leader (head nurse/department leader). Pamphlets will also be distributed with information at the different workplaces. Interested participants with musculoskeletal complaints will then directly book an appointment. An informed consent will be made separately for Study II, and a new one for Study III and IV. According to current rules and regulations regarding responsibility for employees, each work place should maintain regular contact with sick-listed workers and try to include them at work ("Avtale om Inkluderende arbeidsliv"). The additional part will be to fill in questionnaires and agree to a physical examination 4-6 weeks later. Participants will, when included into the RCT in Study III, be asked if they want to take part in the focus group interviews in Study IV. An application for the complete project will be sent to Regional Ethical Committee.

Gender equality and gender perspectives More women than men are working in health care and have a higher percentage of sick-leave, although both gender will be invited to participate. The project will focus on identifying mechanisms for sick-leave absence in a bio-psycho-social perspective, and the gender perspective, both organizational and physical, will be focused on.

6. Communication with users and utilization of results

Communication with users Central users in this project are health workers in the primary health care system and representatives from them have been involved in planning of the project and will continue to be so. The research results will be mediated in meetings with the work group leaders and head nurses and in courses arranged for the employees. The workplace leaders will meet the research team and the appointed course instructors to exchange experience several times throughout the project period.

Dissemination plan The research material will be analyzed and disseminated in articles published in relevant, national and international referee based journals. Furthermore, information will be disseminated by courses and lectures to health workers employed in primary health care facilities, as well as to physiotherapists/manual therapists working in physiotherapy clinics, based on the results of the different studies. It is anticipated that the workplace contacts will continue for workers at risk for becoming sick-listed also after the project has ended, if the study has shown positive results.

ELIGIBILITY:
Inclusion Criteria:

* NSLBP for > 3 months, and reported that their pain was provoked by postures, movement and daily activities.
* Pain intensity measured with a numerical rating scale (NPRS) over the last 14 days >3/10
* Roland Morris Disability Questionnaire (RMDQ) ≥ 7 was necessary to be admitted to the study.
* Ørebro Musculoskeletal Pain Questionnaire-short form (ØMPQ-SF) was used to examine the participants risk profile pre-treatment, and had to be ≥ 30, on a scale from 0-100.

Exclusion Criteria:

* Continuous sick-leave duration ≥ 4 months
* Acute exacerbation of LBP a
* Specific LBP diagnosis - radicular pain, disc herniation, spondylolisthesis, stenosis, Modic changes
* Any low limb surgery in the last 3 months; surgery involving the lumbar spine;
* Pregnancy
* Diagnosed psychiatric disorder
* Active rheumatologic disease, progressive neurological disease
* Serious cardiac or other internal medical condition
* Malignant diseases, acute traumas, infections, or acute vascular catastrophes.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-03; Primary Completion 2016-12 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Sick listing - self reported | Baseline, after 3 months and after 12 months
  Measure if there is a change in self reported sick listing from baseline to after treatment and 12 months follow up

SECONDARY OUTCOMES:
Roland Morris | Baseline, 3 months and 12 months
  self-administered questionnaire with 24 statements about health status, with a score of 0-24, with 0 corresponding to no disability. It has been designed to be completed by patients to assess physical disability due to LBP
Numerical Pain Rating Scale (NPRS) | Baseline, 3 months and 12 months
  Pain intensity in the previous week was the first primary outcome, measured by The NPRS measures pain severity by asking the patient to select a number (from 0 to 10) to represent how severe the pain had been over the last 2 weeks
Hopkins Symptoms Checklist | Baseline, 3 months and 12 months
  A self reported measure of well being. Measure if there is a change in self reported well being from baseline to after treatment and 12 months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Undecided